CLINICAL TRIAL: NCT06739889
Title: Effects of Elongation Longitudinaux Articular Vertebral and Columnar Decoaption Osteo-articulaire Versus Upper Thoracic Mobilization on Forward Head Posture in Upper Cross Syndrome
Brief Title: Effects of ELAVl and CDOA vs Upper Thoracic Mobilization on Forward Head Posture in Upper Cross Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/767
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Cross Syndrome
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group I (Experimental)
  Interventions: Diagnostic Test: Elongation longitudinaux articular vertebral and columnar decoaption osteo-articulaire also known as ELDOA
- Interventional group II (Active Comparator)
  Interventions: Diagnostic Test: upper thoracic mobilization

INTERVENTIONS:
Diagnostic Test: Elongation longitudinaux articular vertebral and columnar decoaption osteo-articulaire also known as ELDOA — ELDOA targtes cervical and upper thoracic spine. ELDOA exercises involves spicific postural holds that improve forward neck posture.The goal of ELDOA is to help reduce stress and increase space in the vertebral joints so that muscles can move freely. The benefits of these stretches include joint mobility, increased fluid absorption in the discs of the spine, flexibility, improved muscle tone, postural alignment, body-mind connection, and coordination. The tension and release created by these stretches helps normalize the posture.
  Arms: Interventional group I
Diagnostic Test: upper thoracic mobilization — Upper thoracic mobilization, often known as joint mobilization, is a common technique in manual therapy. In order to preserve or restore joint mobility, this approach glides and uses distraction on the joint surfaces.
  Arms: Interventional group II

SUMMARY:
This randomized controlled study will examine the patient of forward head posture who suffering with upper cross syndrome. There will be comparison of two treatment methods 1st one is elongation longitudinaux articular vertebral and columnar decoaption osteo-articulaire also known as ELDOA and 2nd is upper thoracic mobilization .

DETAILED DESCRIPTION:
This study includes 42 participants, both male and female, age between 20 to 45. ELDOA target the cervical and upper thoracic spine to improve range of motion, restore normal cervical and thoracic spine alignment and reduce muscle tension. Upper thoracic mobilization improve thoracic spine mobility and enhance cervical spine alignment.

ELIGIBILITY:
Inclusion Criteria:

* Adult between (20 to 45 year) with upper cross syndrome
* CVA angle less than 48-50 degrees.
* No history of spinal injury and fracture
* limited cervical range of motion

Exclusion Criteria:

* Severe spinal degeneration or deformity
* Injury or surgery
* Cervical radiculopathy
* Severe osteoporosis
* Malignancy of upper extremity of thorax
* Obesity

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Tragus to wall test | 12 Months
  Tragus to wall test for forward head posture assessment: normal below 10 centimetres , 10.1- 12 centimetres for mild positive forward head posture,12.1-15 centimetres moderate forward head posture, less than 15 centimetres severe forward head posture.
Craniovertebral angle assess | 12 Months
  Craniovertebral angle assess by web plot digitizer software: normal CVA value 48-50 degree, positive forward head posture less than 48 degree

CONTACTS AND LOCATIONS:
Locations (1):
- Allied hospital, Masjid ismail Rd, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No